CLINICAL TRIAL: NCT06831565
Title: Comparison of Blood Products Required Using Two Different ROTEM Cut-offs Before Invasive Procedures in Cirrhosis and Acute on Chronic Liver Failure (ACLF) Patients With Severe Coagulopathy: A Randomized Controlled Trial
Brief Title: Comparison of Blood Products Required Using Two Different ROTEM Cut-offs Before Invasive Procedures in Cirrhosis and Acute on Chronic Liver Failure (ACLF) Patients With Severe Coagulopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ILBS-ACLF-21
Record Dates: First submitted 2025-01-17; First posted 2025-02-18 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-01

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Cut Off (Active Comparator): EXTEM CT>80sec, CL130<50% FIBTEM- Mcf>8
  Interventions: Diagnostic Test: ROTEM
- High Cut Off (Experimental): EXTEM CT>100sec, CL130<40% FIBTEM- Mcf<6
  Interventions: Diagnostic Test: ROTEM
- On demand (No Intervention): No pre procedure blood products transfusions will be given. Transfusions will be given after the procedure if any bleeding complications occur

INTERVENTIONS:
Diagnostic Test: ROTEM — ROTEM Tests
  Arms: High Cut Off; Low Cut Off

SUMMARY:
Coagulation system in cirrhotics patients is a fragile state , which is rebalanced hemostasis. Standard tests (INR/aPTT) stop measuring at first stage of coagulation ,when the clot first form. VETs measure the whole process such as ROTEM, TEG and comparing these two tests to assess for transfusion of blood products for invasive procedures. . ROTEM provides information both on anti coagulant and procoagulant status where as conventional tests provide only anti coagulant status Invasive procedures can be low risk or high risk or Non surgical vs surgical, Procedure related bleed occurs in 7% of patients with cirrhosis and associated with higher 28 day mortality. MELD, CTP ,AKI , SEPSIS increase the risk of procedure related bleed. Hence for invasive procedures investigator is using relaxing threshold for blood product transfusion in cirrhosis, ACLF patients. As use of ROTEM when compared to conventional tests reduces the need for blood transfusion. Investigator want to proceed with further relaxation of cutoff values of Coagulation parameters and use High cutoff vs low cut off for blood transfusion need.

DETAILED DESCRIPTION:
Aim and Objective - To evaluate the efficacy and safety of relaxed threshold (compared to threshold) for blood product transfusion for invasive procedures in cirrhosis and ACLF patients.

Hypothesis - Relaxing the threshold ( as compared to conventional threshold ) for blood product transfusion will decrease the need for blood products without increase the bleeding complications for invasive procedures in cirrhosis and acute on chronic liver failure patients( ACLF)

Sample size with justification:

Assuming the prevalence rate is 50% (TUSHAR THESIS -yet to be published), that is need of transfusion of blood produtcs in standard cutoff and relaxed cutoff , as according to this study the need in relaxed cut off has been reduced,investigator assumed the need in High cut off group is reduced to 40%, with alpha-5%, power-80%, investigator need to enroll 417 in each group with defaulter of 10% , it decided to have cases that is 934 total Monitoring and assessment: All patients would undergo vital and baseline parameter screening before randomization. Based on randomization investigator will assess the need for transfusion , and complications post procedure , post transfusion if any for a duration of 1month.

Intervention: Patient after screening for all exclusion criteria will be randomized to procedure after or before transfusion of blood products and will be assessed the safety of procedure related bleed and need of intervention post procedure if any

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis and ACLF ( as per definition)
2. Planned to undergo invasive procedures
3. Severe Coagulopathy- INR>2.0 or Platelets <30k or Fibrinogen<100mg/dl .

Exclusion Criteria:

1. Ongoing bleeding
2. Bleeding in past 48 hours before procedure
3. Antiplatelet or anticoagulant therapy ( stopped < 7 days before)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 934 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with reduction in the amount of total components transfused in high cut off ROTEM compared to low cut off ROTEM in cirrhosis and ACLF patients. | Day 28
  High Cutoff defined as need of low blood transfusion products (CT->100sec,MCF<25,CLI30<40%,MCF -FIB<6mm) and Low Cut off defined as (CT ->80sec, MCF<35, CLI30<50%,MCF-FIB<6mm)

SECONDARY OUTCOMES:
Assess the impact of ROTEM on transfusion requirements. | Day 28
  Impact of standard ROTEM on transfusion requirements that is proportion Of FFP, PLATELETS,CRYO, PCC, FIBRINOGEN before procedure in cirrhosis and ACLF patients.
Evaluate the incidence of bleeding events post procedure in Low cutoff. | Day 28
Mortality related with procedural bleeding in both groups. | Day 28
Proportion of the patient requiring procedural based treatment that is number of blood transfusions, angioembolization after post procedural bleed. | Day 28
To compare the rate of transfusion reactions in relaxed ROTEM vs standard ROTEM in cirrhosis and ACLF. | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided